CLINICAL TRIAL: NCT01887275
Title: Medical Ozone Versus Conventional Interferon-α Treatment of Patients With Chronic Hepatitis B -A Control Study to Evaluate The Efficacy And Safety of Ozone-therapy in Chronic Hepatitis B
Brief Title: A Control Study to Evaluate The Efficacy And Safety of Ozone-therapy in Chronic Hepatitis B
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: gyb61641947
Record Dates: First submitted 2013-06-23; First posted 2013-06-26 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2012-10

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic hepatitis B; Medical Ozone; Interferon-α; Efficacy
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- medical ozone therapy with humares (Experimental)
  Interventions: Device: medical ozone therapy with humares
- conventional interferon-α (Active Comparator)
  Interventions: Drug: conventional interferon-α

INTERVENTIONS:
Device: medical ozone therapy with humares — Medical ozone therapy with instrument made in Germany Patients in this group will receive autohemotherapy treatment. First month: ozone concentration: 20µg ~40µg /ml;The second month: 30µg/ml × 100ml oxygen- ozone gas × 100 ml blood;The third month: 20µg/ml × 100ml oxygen- ozone gas× 100 ml blood.
  Other Names: ozone instrument made in Germany: Humares
  Arms: medical ozone therapy with humares
Drug: conventional interferon-α — Patients in the conventional interferon-α treatment group received subcutaneouslly injection of 5 million units of conventional interferon-α in three times per week for at least 24 weeks.
  Arms: conventional interferon-α

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of medical ozone in treatment of chronic hepatitis B patients.

DETAILED DESCRIPTION:
Total of 439 patients with chronic hepatitis B were divided according to patients' intention into two arms. 173 patients in arm I were treated with medical ozone therapy with humares which was made in Germany for at least 12 weeks.266 patients in arm II were treated with conventional interferon-α for at least 24 weeks.Patients in both groups were followed-up for 24 weeks.Virology response, biochemistry response and hepatitis B viral serological response will be studied at 12 weeks after the treatment, at the end of treatment and after 24 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female；
* HBsAg positive for over 6 months；
* ALT over 2×ULN, TBIL less than 80 µmol/L.

Exclusion Criteria:

* Patient has a history of hemorrhagic or hemolysis disease;
* Patient has any history of clinical signs/symptoms of hepatic decompensation or serious metabolic hepatic disease;
* Patient is co-infected with HIV or HCV;
* Patient is treated with anti-virus drug like interferon or nucleoside analogue in recent 6 months;
* Patient is treated with immunosuppressive agent for long time, including patient has a history of organ transplantation;
* Pregnancy;
* Current alcohol or drug abuse;
* Difficulty to draw blood through veins;
* Patient has a history of carcinoma, or finding suggestive of possible hepatocellular carcinoma (HCC), or AFP over than 100ng/ml;
* Patient has a history of any severe physical disease such as cardio-vascular, kidney events, hyperthyroidism or serious electrolyte disturbance;
* Patient is enrolled in any other clinical trials.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 439 (Actual)
Dates: Start 2010-03; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
HBV DNA | up to 77 weeks
  To demonstrate the percentage of patients achieving HBV DNA<1000copies/mL

SECONDARY OUTCOMES:
HBeAg | up to 77 weeks
  Percentage of patients with HBeAg loss and HBeAg seroconversion in patients with HBeAg positive at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: yabing guo, professor, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Guangzhou, Guangdong, China